CLINICAL TRIAL: NCT02153528
Title: Optimization of the TB Treatment Regimen Cascade
Acronym: OneRIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Damien Foundation (Other)
Collaborators: National TB control Programme Bangladesh (Other); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OneRIF
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Bangladesh; Rimfapicin
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard TB treatment (Active Comparator): Standard regimen for TB treatment according to guidelines of the International Union against Tuberculosis and Lung Disease
  Interventions: Drug: Standard TB treatment
- double rimfampicin (Experimental): 2HREZ/4HR Cat. 1, modified by using double dose rifampicin throughout
  Interventions: Drug: double rimfampicin

INTERVENTIONS:
Drug: double rimfampicin — Compared to standard regimen dosing of rifampicin is doubled, while standard dose isoniazid, pyrazinamide and ethambutol are maintained
  Other Names: Intervention arm
  Arms: double rimfampicin
Drug: Standard TB treatment — Standard regimen for TB treatment according to guidelines of the International Union against Tuberculosis and Lung Disease
  Other Names: Control arm
  Arms: Standard TB treatment

SUMMARY:
- Hypothesis: Double dose rifampicin together with earlier monitoring of sputum conversion using vital staining reduces unfavorable outcome of Cat. 1 first-line TB treatment without excess serious toxicity, and allows early switch to specific treatment of MDR-TB without using Cat. 2 retreatment regimen

- General study design: This open label, randomised clinical trial is intended as a pilot study on the efficacy and safety of high-dose rifampicin and feasibility and added value of auramine and/or FDA vital staining sputum smear after 2 weeks of intensive treatment phase. If this proof-of-concept study provides substantial indication of benefit without indication of excess toxicity, the data from the study will be used to design a larger scale, cluster-randomized study. The aim of this cluster randomised study would be to provide definite proof of the benefit of the intervention on adverse treatment outcomes and lack of excess toxicity associated with high dose rifampicin. In addition, the cluster-randomized study would provide a more precise assessment of the suppression and prevention of (acquired) resistance endpoints.

An interim analysis is thus planned at the time the last recruited patient finishes treatment, i.e. about 9 months after the end of recruitment. It will focus on assessment of drug toxicity versus suggested benefits of the intervention. This analysis will be primarily performed for the go/no-go decision and design considerations for the cluster-randomized trial. The decision on proceeding to the cluster randomized study will be based on the absence of excess toxicity, a trend toward a reduction of unfavourable outcomes (excluding relapse), and possible favourable effects on initially present low-resistance mutations / mutations acquired during treatment. It will also allow to adapt the design of the larger study particularly regarding the algorithm for resistance screening, and whether or not treatment shortening could be justified with rapid initial conversion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with smear-positive pulmonary TB
* 15 years or older
* Able and willing to provide written informed consent

Exclusion Criteria:

* contacts of MDR-TB patients and other MDR-TB suspects diagnosed with resistance on rapid DST for rifampicin performed prior to start of treatment according to NTP guidelines
* smear-negative pulmonary and extra-pulmonary TB cases
* patients in need of hospitalization because of very bad general condition or complications
* patients with clinically active liver disease, for the study defined as jaundice confirmed by a local Medical Officer (Government)
* any known HIV-positive patient (although none are expected)
* any patient with known hepatitis B or C infection
* pregnant women; in addition, patients in the intervention arm who become pregnant during treatment will be switched to the control arm

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2014-11; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aung Kya Jai Maug, MD, Principal Investigator — Damien Foundation Bangladesh
Locations (1):
- Damien Foundation Bangladesh TB project in Greater Mymensingh district (8 selected clinics), Dhaka, Greater Mymensingh District, Bangladesh

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard TB Treatment | Double Rimfampicin
Started | 348 | 353
Completed | 348 | 353
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 3 subjects (1 from intervention arm and 2 from control arm) were excluded from the baseline population because they were infected with Non-TB-Mycobacteria (NTM).
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard TB Treatment | Double Rimfampicin | Total
Number analyzed (Participants) | 346 | 352 | 698
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [28 to 55] | 45 [27.5 to 55] | 44 [28.0 to 55.0]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 251 | 260 | 511
  Female | 95 | 92 | 187
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Median (Inter-Quartile Range); unit: kg] | 41 [37 to 46] | 42 [36 to 46] | 41.5 [36 to 46]
Height [Median (Inter-Quartile Range); unit: cm] | 159 [153 to 165] | 158 [152 to 164] | 159 [152 to 164]
Temperature [Median (Inter-Quartile Range); unit: °F] | 99.1 [98.3 to 100.2] | 99.2 [98.5 to 100.0] | 99.2 [98.4 to 100.2]
Direct smear auramine [Median (Inter-Quartile Range); unit: Acid Fast Bacilli/field] — 200x magnification
  Acid Fast Bacilli/field | 98 [7.0 to 550.0] | 90.0 [7.0 to 500] | 93.3 [7.0 to 525.0]
Intervention smear auramine [Median (Inter-Quartile Range); unit: AFB/field] — 200x magnification
  AFB/field | NA [NA to NA] — This was only assessed for the intervention arm (double rifampicin). | 100.0 [8.0 to 575.0] | 100.0 [8.0 to 575.0]
Intervention smear FDA [Median (Inter-Quartile Range); unit: number of AFB] — 200x magnification
  number of AFB | NA [NA to NA] — Only assessed in het intervention arm (double rifampicin). | 10.0 [0.5 to 79.5] | 10.0 [0.5 to 79.5]
ALT [Median (Inter-Quartile Range); unit: IU/L] | 20 [14 to 33] | 20 [15 to 29.5] | 20 [15 to 31]
New case of TB [Count of Participants; unit: Participants]
  No | 20 | 29 | 49
  Yes | 326 | 323 | 649
Diabetes [Count of Participants; unit: Participants]
  No | 331 | 335 | 666
  Yes | 15 | 17 | 32
Liver problems [Count of Participants; unit: Participants]
  No | 346 | 351 | 697
  Yes | 0 | 1 | 1
Kidney problems [Count of Participants; unit: Participants]
  No | 346 | 351 | 697
  Yes | 0 | 1 | 1
Lung/Heart problems [Count of Participants; unit: Participants]
  No | 344 | 349 | 693
  Yes | 2 | 3 | 5
Sign of Hepatitis [Count of Participants; unit: Participants]
  No | 346 | 352 | 698
  Yes | 0 | 0 | 0
Cough [Count of Participants; unit: Participants]
  No | 1 | 1 | 2
  Yes | 345 | 351 | 696

OUTCOME MEASURES:

1. Primary Outcome: Tuberculose Treatment Outcome
Description: Following current WHO guidelines, an adverse treatment outcome is defined as any occurrence of the following:
  * Relapse: Cured previously from TB or completed treatment for TB and now having bacteriologically positive sputum for TB (at 12 months follow-up or at an earlier time point)
  * Default: The patient whose treatment was interrupted for ≥ 2 consecutive months.
  * Failure: Sputum positive for TB at 5 months or later during treatment. In line with current WHO recommendations, patients detected with MDR-TB or rifampicin resistance before this or another outcome applies and switched to the MDR-TB regimen will be excluded from the outcome analysis.18 Failure will also be declared if the regimen has to be changed for at least 2 drugs due to adverse events.
  * Death: All-cause mortality between case registration and end of TB treatment (related or not to TB or TB treatment)
Time Frame: 12 months after end of treatment
Population: Intention-to-treat analysis. Additional 4 subjects were removed from the ITT analysis because they switched to MDR regimen (3 in control arm, 1 in intervention arm). 4 subjects (intervention arm) were removed from the ITT analysis because they were enrolled twice.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 343 | 347
Participants
  Default | 8 | 8
  Died | 11 | 5
  Failure | 8 | 12
  Completed | 6 | 3
  Cured | 310 | 319

2. Primary Outcome: Number of Participants Who Develop Liver Toxicity
Description: Grade 3-4 Liver Toxicity following NIH common toxicity criteria (CTC), including transaminase increases to >5-20 ULN (grade 3), or > 20 ULN (grade 4)
Time Frame: until month eight
Population: One participant was allocated to double rifampicin arm but received standard TB treatment, and was analysed in the standard TB treatment arm.Two participants were deleted from analysis because they had grade 3 liver toxicity at baseline and 6 participants were deleted because they did not have any follow-up ALT values.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 343 | 350
Participants | 7 | 3

3. Secondary Outcome: High-level Rifampicin Resistant TB Adverse Treatment Outcomes
Description: To assess whether the study regimen also cures high-level rifampicin resistant TB. Adverse treatment outcomes will be described and compared among treatment groups in subgroups defined by initial rifampicin resistance mutations (performed in all patients) detected.
Time Frame: 12 months after end of TB treatment
Population: ITT analysis population. Compared to analysis population of primary objective - TB treatment outcome, 24 subjects were excluded from this analysis due to missing or negative sequencing results (8 in control group, 16 in intervention group).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 335 | 331
Participants
  Rif-sensitive with adverse treatment outcome | 52 | 40
  Rif-sensitive cured/completed without relapse | 281 | 290
  Rif-resistant with adverse treatment outcome | 0 | 0
  Rif-resistant cured/completed without relapse | 2 | 1

4. Secondary Outcome: Number of Initial Resistant TB Cases Who Switched to MDR-TB Treatment or Were Cured
Description: To assess the effectiveness of FDA vital staining versus fever screening for early switch of non-responding rifampicin resistant TB to MDR-TB treatment
Time Frame: at two weeks of treatment
Population: 7 initial resistant cases (5 in control group and 2 in intervention group).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 5 | 2
Participants | 5 | 2

5. Secondary Outcome: the Negative Predictive Value of Conversion at 2 Weeks for Relapse.
Description: The Negative Predictive value (and 95% CI) of conversion in the intervention arm will be estimated as the % of relapses among those with a minimum 1 log decline in the number of AFB, or who are already negative or only scanty positive on AFB smear (auramine or FDA).
Time Frame: at 2 weeks of treatment
Population: ITT analysis. This analysis only includes participants in the intervention arm who are negative on auramine smear resp. FDA smear at 2 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Double Rifampicin Arm Negative on Auramine Smear: This outcome is only calculated for the intervention arm.
- Double Rifampicin Group Negative on FDA Smear: This outcome is only analysed for the intervention arm.
Arm/Group | Double Rifampicin Arm Negative on Auramine Smear | Double Rifampicin Group Negative on FDA Smear
Number analyzed (Participants) | 91 | 193
Participants | 0 | 0

6. Secondary Outcome: Proportion of Acquired Rifampicin Resistance Among Failures and Relapses
Description: number of failure / relapse cases without mutation detected at diagnosis as the denominator and comparing intervention and control arms.
Time Frame: 12 months after end of TB treatment
Population: ITT analysis. This analysis only includes failure / relapse cases without mutation detected at diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 8 | 12
Participants | 0 | 0

7. Secondary Outcome: Area Under the Curve of Auramine Resp. FDA at 2 Weeks to Predict Adverse Treatment Outcome at 1 Year After Treatment Completion
Description: Area under the ROC curve (AUC) to predict adverse treatment outcome. The X-axis represents the 1-specificity, the Y-axis represents sensitivity. The AUC is estimated with 95% confidence interval.
Time Frame: Auramine/FDA at 2 weeks and adverse treatment outcome 1 year after treatment completion
Measure: Number (95% Confidence Interval); unit: no unit is used for AUROC
Arm/Group | Double Rifampicin Arm Negative on Auramine Smear | Double Rifampicin Group Negative on FDA Smear
Number analyzed (Participants) | 344 | 344
no unit is used for AUROC | 0.52 [0.42 to 0.61] | 0.54 [0.45 to 0.63]

8. Secondary Outcome: Weight Gain
Description: Weight gain from baseline until end-of-treatment comparison between both treatment arms.
Time Frame: until end of treatment (month eight)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 320 | 331
kg | 2.93 (2.44) | 2.79 (2.44)

9. Secondary Outcome: Fever Resolution
Description: Comparison of fever resolution after 2 weeks of treatment between both treatment arms.
Time Frame: after 2 weeks of treatment
Population: Total of participants with fever at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard TB Treatment | Double Rimfampicin
Number analyzed (Participants) | 82 | 72
Participants | 81 | 71

ADVERSE EVENTS:
Time Frame: Serious adverse events are recorded until end of treatment (up to 8 months). No (non-serious) adverse events are recorded in this trial.
Arm/Group | Standard TB Treatment | Double Rimfampicin
All-Cause Mortality (participants affected / at risk) | 17/348 | 12/353
Serious Adverse Events (participants affected / at risk) | 24/348 | 13/353
Other Adverse Events (participants affected / at risk) | 0/348 | 0/353
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard TB Treatment (N=348) | Double Rimfampicin (N=353)
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 4 | 5
Alanine aminotransferase increased (Investigations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Victim of homicide (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT02153528/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT02153528/SAP_001.pdf